CLINICAL TRIAL: NCT03587168
Title: The Reliability, Validity, and Responsiveness of the Timed 360° Turn Test in Patients With Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Fatih Söke, Research Assistant, Gazi University
Other Study IDs: 441
Record Dates: First submitted 2018-07-03; First posted 2018-07-16 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; The Timed 360° Turn Test; Validity; Reliability
MeSH Terms: conditions — Parkinson Disease | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Parkinson's Disease: Patients with Parkinson's Disease Parkinson's Disease (Hoehn and Yahr stage 1-4)
  Interventions: Other: the timed 360° turn test; Other: Berg Balance Scale; Other: Four Square Step Test; Other: Functional Reach Test; Other: Trunk Impairment Scale; Other: Timed Up and Go Test; Other: Hoehn and Yahr Scale; Other: Unified Parkinson's Disease Rating Scale
- Healthy Controls: Healthy People
  Interventions: Other: the timed 360° turn test

INTERVENTIONS:
Other: the timed 360° turn test — Turning ability is assessed by using the timed 360° turn test.
Other: Berg Balance Scale — Functional balance is assessed by using the Berg Balance Scale.
  Groups: Patients with Parkinson's Disease
Other: Four Square Step Test — The Four Square Step Test measures dynamic balance.
  Groups: Patients with Parkinson's Disease
Other: Functional Reach Test — The Functional Reach Test assesses limits of stability.
  Groups: Patients with Parkinson's Disease
Other: Trunk Impairment Scale — Trunk performance is assessed by using the trunk impairment scale.
  Groups: Patients with Parkinson's Disease
Other: Timed Up and Go Test — Functional mobility is assessed by using the timed up and go test.
  Groups: Patients with Parkinson's Disease
Other: Hoehn and Yahr Scale — Disease stage is assessed by the Hoehn and Yahr Scale.
  Groups: Patients with Parkinson's Disease
Other: Unified Parkinson's Disease Rating Scale — The Unified Parkinson's Disease Rating Scale assesses disease severity.
  Groups: Patients with Parkinson's Disease

SUMMARY:
Difficulty in turning is common after Parkinson's Disease. Patients with Parkinson's Disease take a greater number of steps, longer duration, narrower base of support in turning. Thus, turning ability is systematically investigated in Parkinson's Disease. The aim of this study to invastigate reliability, validity, and responsiveness of the timed 360° turn test in Patients with Parkinson's Disease.

DETAILED DESCRIPTION:
At baseline, the timed 360° turn test, Unified Parkinson's Disease Rating Scale, Hoehn and Yahr Scale, Berg Balance Scale, Functional Reach Test, Timed Up and Go Test, Four Square Step Test and Trunk Impairment Scale was applied to the patients with Parkinson's Disease when the patients were "on" period. The timed 360° turn test was repeated after seven days from the first application when patients with Parkinson's Disease were "on" period to evaluate its reliability.

ELIGIBILITY:
Inclusion Criteria:

* at least 40 years of age,
* neurologist-diagnosed Parkinson's Disease
* Hoehn & Yahr (H&Y) stages 1 to 4,
* were able to walk 10 m with or without aids

Exclusion Criteria:

* visual, auditory, and orientational problems affecting study results
* orthopedic problems affecting walking,
* other neurologic conditions, cardiovascular, musculuskeletal, and vestibular disease

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's Disease who apply to the Gazi University, Department of Physiotherapy and Rehabilitation will be invited to this study.
Sampling Method: Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2018-07-20 (Actual); Primary Completion 2018-08-10 (Actual); Study Completion 2018-08-20 (Actual)

PRIMARY OUTCOMES:
The timed 360° turn test | 10 seconds
  Turning ability is assessed by using the timed 360° turn test. In the timed 360° turn test, a piece of colored tape is placed on the floor to mark the starting position. Each subject was required to stand with arms by his/her side and feet comfortably apart and pointing to the tape. Timing was started from the word "go" and stopped when subject's shoulders were facing forward again. The time taken to complete the turn was recorded (in seconds) by a stopwatch.

SECONDARY OUTCOMES:
Berg Balance Scale | 15 minutes
  Functional balance is assessed by using the Berg Balance Scale. During the test, participants are asked to perform 14 tasks frequently used in daily life activities. Each item is scored between 0 (unable to perform the task) and 4 (task is performed independently) according to the ability of the person while performing the task. The highest possible score is 56 points. A higher score indicates better balance.
Trunk Impairment Scale | 20 minutes
  Trunk performance is assessed by using the trunk impairment scale. The Trunk Impairment Scale consists of three subscales: static sitting balance, dynamic sitting balance and co-ordination. A higher score indicating a better performance.
Functional Reach Test | 15 seconds
  The Functional Reach Test assesses balance by measuring the limits while the patient reaches forwards as far as possible, having the arms in 90° flexion and without lifting the heels off the floor.
Four Square Step Test | 15 seconds
  The Four Square Step Test measures dynamic balance and clinically assesses the person's ability to step over objects forward, sideways, and backward. A square was formed by 4 canes resting flat on the floor. The participants were instructed to try and complete the sequence as fast as possible without touching the canes with both feet, making contact with the floor in each square.
Timed Up and Go Test | 10 seconds
  Functional mobility is assessed by using the timed up and go test. The timed up and go test measures the time that a patient needs to stand up from a chair, walk a 3-m distance, come back and sit back on the chair.
Hoehn and Yahr Scale | 1 minutes
  Disease stage is assessed by the Hoehn and Yahr Scale. The Hoehn and Yahr scale is a commonly used diagnostic tool for quantifying the progression of Parkinson's Disease symptoms. Stages range from 0 (no signs of disease) to 5 (requiring a wheelchair, or bedridden unless assisted).
Unified Parkinson's Disease Rating Scale | 15 minutes
  The Unified Parkinson's Disease Rating Scale is increasingly used as a gold standard reference scale and includes four components (Part I, Mentation, Behavior and Mood; Part II, Activities of Daily Living; Part III, Motor;Part IV, Complications). A lower score indicates lower disease severity.

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Söke, Principal Investigator — Gazi University
Locations (1):
- Fatih Söke, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schenkman M, Cutson TM, Kuchibhatla M, Chandler J, Pieper C. Reliability of impairment and physical performance measures for persons with Parkinson's disease. Phys Ther. 1997 Jan;77(1):19-27. doi: 10.1093/ptj/77.1.19. PMID 8996460
- [Background] Stack E, Ashburn A. Dysfunctional turning in Parkinson's disease. Disabil Rehabil. 2008;30(16):1222-9. doi: 10.1080/09638280701829938. PMID 18608364
- [Background] Kluger BM, Brown RP, Aerts S, Schenkman M. Determinants of objectively measured physical functional performance in early to mid-stage Parkinson disease. PM R. 2014 Nov;6(11):992-8. doi: 10.1016/j.pmrj.2014.05.013. Epub 2014 May 28. PMID 24880056
- [Background] Stack EL, Ashburn AM, Jupp KE. Strategies used by people with Parkinson's disease who report difficulty turning. Parkinsonism Relat Disord. 2006 Mar;12(2):87-92. doi: 10.1016/j.parkreldis.2005.08.008. Epub 2005 Dec 9. PMID 16338159
- [Background] Shiu CH, Ng SS, Kwong PW, Liu TW, Tam EW, Fong SS. Timed 360 degrees Turn Test for Assessing People With Chronic Stroke. Arch Phys Med Rehabil. 2016 Apr;97(4):536-544. doi: 10.1016/j.apmr.2015.11.010. Epub 2015 Dec 13. PMID 26694578
- [Background] Giladi N, McMahon D, Przedborski S, Flaster E, Guillory S, Kostic V, Fahn S. Motor blocks in Parkinson's disease. Neurology. 1992 Feb;42(2):333-9. doi: 10.1212/wnl.42.2.333. PMID 1736161